CLINICAL TRIAL: NCT04089501
Title: The Role of the Pregnane X Receptor (PXR) in Indole Signaling and Intestinal Permeability in Inflammatory Bowel Disease
Status: Completed | Type: Observational
Sponsor: Albert Einstein College of Medicine (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Sridhar Mani, Principal Investigator, Albert Einstein College of Medicine
Other Study IDs: 2015-4465; 3R01CA127231 (NIH); 5R01CA161879 (NIH)
Record Dates: First submitted 2019-09-12; First posted 2019-09-13 (Actual); Last update posted 2019-09-16 (Actual); Status verified 2019-09

CONDITIONS: Inflammatory Bowel Diseases
MeSH Terms: conditions — Inflammatory Bowel Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Tissue, Stool
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Inflammatory Bowel Disease (IBD): Subjects will be asked to provide a stool sample (if no colonoscopy is to be performed) or if clinically indicated, a colonoscopy will be performed per standard medical routine. During colonoscopy, stool will be collected for analysis and 3 additional biopsies will be taken each from the ileum and colon for research purposes. Alternatively, subjects who are undergoing intestinal and/or colonic resection will provide stool prior to surgery and a portion of their pathology specimens will be used for research purposes following complete pathologic evaluation.
  Interventions: Diagnostic Test: Stool collection; Diagnostic Test: Biopsy collection
- Subjects not affected by IBD (Control Group): Results of subjects with IBD will be compared to subjects in the control group.
  Interventions: Diagnostic Test: Stool collection; Diagnostic Test: Biopsy collection

INTERVENTIONS:
Diagnostic Test: Stool collection — Stool will be collected from subjects who have been diagnosed with IBD or whom small intestinal, colonic or ileocolonic and have signed consent for the control group. Stool will be self-collected or through routine colonoscopy procedure.
Diagnostic Test: Biopsy collection — 3 additional biopsies (for research purposes) will be taken from patients who undergo colonoscopy as per standard of care

SUMMARY:
The goal of this study is to better understand the mechanisms responsible for the development of and the severity of Inflammatory Bowel Disease (IBD), such as Crohn's Disease and Ulcerative Colitis, which cause inflammation of the gut as well as potentially affecting other areas of the body

DETAILED DESCRIPTION:
Based on promising preliminary data, the study will characterize the claim that PXR signaling serves as a key mechanistic link between the host environment and the innate immune system in the gut. It is widely believed that one cause of IBD stems from abnormal sensing of commensal bacteria. The research will shed light on the molecular mechanisms used by gut barrier epithelial cells in sensing commensals and regulating inflammatory responses in the gut. This will provide a new mechanism towards which more mechanisms derived probiotics could be used to abrogate intestinal inflammation. It is hoped that these agents would eventually serve as non-toxic alternatives or adjuncts to currently available therapeutics for IBD. The research protocol will involve the collection of feces, either by self-collection or through colonoscopic washing.

ELIGIBILITY:
Inclusion Criteria:

i) IBD patients

* Patients aged 18-65 with a diagnosis of Crohn's disease, ulcerative colitis, or indeterminate colitis
* Willing and able to consent to participation in study
* In order to enroll in complete study, a clear indication for colonoscopy must be present. If colonoscopy is not indicated, patients may elect to participate by providing a stool specimen without undergoing colonoscopy.
* IBD patients with a clinical recommendation for small intestinal, colonic, or ileocolonic resection

ii) Control patients

* Patients aged 18-65 with no diagnosis of inflammatory bowel disease being seen in the gastroenterology practice for the following indications

  * Screening colonoscopy
  * Iron deficiency anemia
  * Rectal bleeding
  * Esophageal reflux (colonoscopy only would be done if indicated for other reasons)
  * Diarrhea (with exclusion of inflammatory bowel disease)
* Patients with no diagnosis of inflammatory bowel disease being seen in the surgery practice in whom small intestinal, colonic, or ileocolonic resection is recommended

iii) Pre-existing specimens from IBD patients

• Pre-existing specimens from the IBD patient tissue biobank of Dr. Gitit Tomer will also be analyzed. Only patient samples from patients who have provided informed written consent for use in future studies on the consent form for the pediatric IBD tissue biobank will be utilized in this study. Such patient specimens will be assigned a unique study identifier and the data will be stored as indicated below. There are currently 38 patients within this biobank, of which all 38 provided consent for use of the specimens in future studies. Specimens include both ileal and colonic biopsies, ileal and colonic fecal aspirates, and serum.

iv) Pediatric IBD patients

* Patients aged 0-22 with a diagnosis of Crohn's disease, ulcerative colitis, indeterminate colitis, or a family history of IBD
* Willing and able to consent to participation in study, or a parent or guardian provides written consent for participation
* In order to enroll in the complete study, a clear indication for colonoscopy and biopsy must be present. If colonoscopy is not indicated, patients may elect to participate by providing a stool specimen without undergoing colonoscopy.
* Pediatric IBD patients with a clinical recommendation for small intestinal, colonic, or ileocolonic resection

Exclusion Criteria:

* Unwilling or unable to provide consent
* Presence of comorbid systemic inflammatory disorders such as rheumatoid arthritis, sarcoidosis, psoriasis, multiple sclerosis, advanced or decompensated heart failure, cirrhosis, or morbid obesity (Body mass index (BMI) over 40)
* Irritable bowel syndrome
* Bowel obstruction
* Contraindication to colonoscopy or biopsies
* Cancer or malignancy within 12 months

Max Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects belonging to the target population, (i.e., Diagnosed with IBD, specifically Crohn's disease, ulcerative colitis, or indeterminate colitis and patients with no diagnosis of IBD in whom small intestinal, colonic, or ileocolonic resection is recommended.
Sampling Method: Non-Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2015-02-25 (Actual); Primary Completion 2019-05-02 (Actual); Study Completion 2019-05-02 (Actual)

PRIMARY OUTCOMES:
Analysis of molecular studies in subjects with and without IBD | Up to 5 years
  We will measure and analyze RNA and protein levels of cytokines, junctional protein expression, PXR (pregnane X receptor) and TLRs (toll-like receptors) in tissues and perform intestinal permeability studies in subjects with and without IBD.
Assays for biofilm and phage | Up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Sridhar Mani, MD, Principal Investigator — Albert Einstein College of Medicine
Locations (1):
- Montefiore Medical Center, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No